CLINICAL TRIAL: NCT04845386
Title: A Comparison of Neuromuscular Transmission in the Arm and Hand Muscles With Alternative Muscles Such as the Lower Leg Muscles and the Corrugator Supercilii During General Anesthesia
Brief Title: : A Comparison of Neuromuscular Transmission in the Muscles During General Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Collaborators: Regional Specialized Hospital in Olsztyn (Unknown)
Responsible Party: Principal Investigator, Radkowski Paweł MD PhD, Principal Investigator, University of Warmia and Mazury in Olsztyn
Other Study IDs: Mivacron 2021
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Neuromuscular Blockade
Keywords: TOF Cuff; TOF Scan; Neuromuscular transmission; corrugator supercilii; Mivacurium; adductor pollicis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TOF Cuff on arm and TOF Scan on corrugator supercilii: Patients undergoing surgery with intubation and receiving a intubation dose of mivacurium (0.2 mg/kg) and repeated dose of mivacurium (2mg) depending of needing under, routine gas anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: TOF Cuff on arm; Device: TOF Scan on corrugator supercilii
- TOF Cuff on lower leg and TOF Scan on adductor pollicis: Patients undergoing surgery with intubation and receiving a intubation dose of mivacurium (0.2 mg/kg) and repeated dose of mivacurium (2mg) depending of needing under, routine gas anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: TOF Cuff on lower leg; Device: TOF Scan on adductor pollicis
- TOF Scan on adductor pollicis and TOF Scan on toe: Patients undergoing surgery with intubation and receiving a intubation dose of mivacurium (0.2 mg/kg) and repeated dose of mivacurium (2mg) depending of needing under, routine gas anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: TOF Scan on toe; Device: TOF Scan on adductor pollicis
- TOF Scan on adductor pollicis and TOF Cuff on arm: Patients undergoing surgery with intubation and receiving a intubation dose of mivacurium (0.2 mg/kg) and repeated dose of mivacurium (2mg) depending of needing under, routine gas anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: TOF Cuff on arm; Device: TOF Scan on adductor pollicis
- TOF Scan on adductor pollicis and TOF Scan on corrugator supercilii: Patients undergoing surgery with intubation and receiving a intubation dose of mivacurium (0.2 mg/kg) and repeated dose of mivacurium (2mg) depending of needing under, routine gas anesthesia will have monitoring of neuromuscular block with two monitors simultaneously.
  Interventions: Device: TOF Scan on adductor pollicis; Device: TOF Scan on corrugator supercilii

INTERVENTIONS:
Device: TOF Cuff on arm — The TOF Cuff will be installed on one arm in opposite of TOF Scan. After intubation dose of mivacurium continuous monitoring of neuromuscular block started until complete recovery of neuromuscular block.
  Groups: TOF Cuff on arm and TOF Scan on corrugator supercilii; TOF Scan on adductor pollicis and TOF Cuff on arm
Device: TOF Cuff on lower leg — The TOF Cuff will be installed on one lower leg. After intubation dose of mivacurium continuous monitoring of neuromuscular block started until complete recovery of neuromuscular block.
  Groups: TOF Cuff on lower leg and TOF Scan on adductor pollicis
Device: TOF Scan on toe — The TOF Scan will be installed on hallux . After intubation dose of mivacurium continuous monitoring of neuromuscular block started until complete recovery of neuromuscular block.
  Groups: TOF Scan on adductor pollicis and TOF Scan on toe
Device: TOF Scan on adductor pollicis — The TOF Scan will be installed on Thumb. After intubation dose of mivacurium continuous monitoring of neuromuscular block started until complete recovery of neuromuscular block.
  Groups: TOF Cuff on lower leg and TOF Scan on adductor pollicis; TOF Scan on adductor pollicis and TOF Cuff on arm; TOF Scan on adductor pollicis and TOF Scan on corrugator supercilii; TOF Scan on adductor pollicis and TOF Scan on toe
Device: TOF Scan on corrugator supercilii — The TOF Scan will be installed on corrugator supercilii. After intubation dose of mivacurium continuous monitoring of neuromuscular block started until complete recovery of neuromuscular block.
  Groups: TOF Cuff on arm and TOF Scan on corrugator supercilii; TOF Scan on adductor pollicis and TOF Scan on corrugator supercilii

SUMMARY:
The investigators want to compare new muscle relaxation monitoring, TOF-Cuff and TOF-Scan, during general anesthesia. Standard monitoring is using thumb, however it can't be use on every patient. Alternative can be eyebrow muscle or foot muscle.

There is only few old study that compares this muscle and used mivacurium. The study aims to compare TOF-Cuff and TOF-Scan with different sensor and use mivacurium.

DETAILED DESCRIPTION:
In our research in addition to the standard intraoperative monitoring, which includes the assessment of ECG and saturation, the investigators would like to estimate muscle relaxation by using two different methods: a TOF-Cuff which additionally allows to measure inoperative blood pressure and TOF-Scan with different sensor. Our aim is to compare two different methods of muscle relaxation monitoring in patients who will administer muscle relaxant - mivacurium. After receiving painkillers and hypnotics, when the patient is falling asleep, the standard dose of mivacurium 0.2 mg / kg body weight will be administered. Then, painless simultaneous stimulation with TOF-Cuff and TOF-Scan devices will begin. Until intubation, measurements will be made in every 30 seconds and then every 5 minutes until extubation. Extubation will take place according to the guidelines when the TOF-Cuff measurement on the arm is greater than 0.9 - this is the value at which the patient is considered ready to start breathing on his own. The following will be documented: the initiation of drug administration, intubation, possible repeated doses of mivacurium 2 mg, antagonization, extubation, possible side effects (e.g., transient cardiac disturbances, reddening of the skin, lowering blood pressure, bronchospasm, erythema, urticaria) and technical problems.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* ASA classification I,II,III
* Elective surgery
* BMI(body mass index) 17-35
* Surgery in the supine position
* Informed consent of the patient

Exclusion Criteria:

* Pregnancy and breastfeeding
* Urgent indications for surgery
* ASA classification >III
* Neuromuscular diseases
* Polyneuropathy
* Diabetes
* Drug addiction
* Family history of malignant hyperthermia
* Allergic to propofol, fentanyl or mivacurium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study will take patients qualified to the elective surgery
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Onset time | 1 to 10 minutes
  Time in seconds from start of injection of mivacurium until emergence of TOF ratio of 0%. TOF = Train of Four
Total recovery time of neuromuscular block | 30 to 500 minutes
  The total recovery time, i.e. total duration of the neuromuscular block is defined as the time in minutes from start of injection of mivacurium until a normalized TOF ratio of 90%

SECONDARY OUTCOMES:
Time to repeated dose | 5 to 200 minutes
  Time in minuted from TOF ratio 0% to repeated dose

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinical Ward, Regional Specialized Hospital, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radkowski P, Rusc J, Keska M, Onichimowski D. Comparison of TOF scan neuromuscular monitoring on adductor pollicis vs. corrugator supercilii and flexor hallucis brevis. Sci Rep. 2025 Jul 14;15(1):25426. doi: 10.1038/s41598-025-11259-5. PMID 40659829